CLINICAL TRIAL: NCT00036179
Title: An Open-Label, Non-Comparative Study of FK463 in the Treatment of Candidemia or Invasive Candidiasis
Brief Title: Study of FK463 in the Treatment of Candidemia or Invasive Candidiasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FG463-21-02; 98-0-047
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2015-06

CONDITIONS: Candidiasis
Keywords: Candidemia; Anti-Fungal
MeSH Terms: conditions — Candidiasis; Candidemia | interventions — Micafungin

INTERVENTIONS:
Drug: FK463

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of FK463 in the treatment of patients with confirmed candidemia or invasive candidiasis.

DETAILED DESCRIPTION:
This will be an open-label, non-comparative study of intravenous FK463. Enrollment will include at least 100 patients evaluable for efficacy.

ELIGIBILITY:
Inclusion Criteria

* Has Candidemia or invasive candidiasis documented by typical clinical signs and symptoms and confirmed by fungal culture or histologic confirmation

Exclusion Criteria

* Has abnormal liver test parameters, e.g., AST or ALT > 10 times upper limit of normal
* Has life expectancy judged to be less than 5 days
* De novo patients who have received a systemic antifungal agent for the treatment of this episode of candidemia or invasive candidiasis for more than 48 hours prior to the first dose of FK463; or efficacy failure patients who have received =< 5 days of prior systemic antifungal therapy for the treatment of this episode of candidemia or invasive candidiasis
* Require treatment with topical or systemic antifungal agents for conditions other than candidemia or invasive candidiasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 1999-02-27 (Actual); Primary Completion 2002-01-27 (Actual); Study Completion 2002-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- Austria (2):
  - Medizinische Univ.-Klinik, Graz
  - Krankenhaus Elisabethinen Linz, Linz
- France (4):
  - Hopital Henri Mondor, Dervice d'Hematologie Clinique, Créteil
  - Hotel Dieu, Service d"Hematologie, Nantes
  - Hopital Saint Louis, Service D'Hematologie/Greffe de Moelle, Paris
  - Hopital Necker Enfants Malades, Service d"Hematologie, Paris
- Germany (7):
  - Johann Wolfgang Goethe Universitat, Medizinische Klinik III, Frankfurt
  - Westpfalz Krankenhaus, Kaiserslautern
  - Medizinische Klinik und Poliklinik II, Abt. Hamatologie und Onkologie, Leipzig
  - Klinikum der Stadt, Medizinische Klinik A, Ludwigshafen
  - Uniklinik Mainz, III. Medizinische Klinik, Mainz
  - LMU Munchen, Hamatopoetische Zell - Transplantation, München
  - Universitat Wurzburg, Institut fur Molekulare und Infectionsbiologie, Würzburg
- Italy (2):
  - Nationale Institute for Cancer Research, Genova
  - Ospedale Niguarda-Ca Granda, Dept. of Internal Medicine Padiglione Brera, Milan
- Institute of Haematology and Blood Transfusion, Warsaw, Poland
- Spain (3):
  - Hospital Clinic I Provencial, Servicio Enfermadades Infecciosas, Barcelona
  - Hospital Gregorio Maranon, Servicio de Enfermadades Infecciosas, Madrid
  - Hospital Doce de Octubre, Servicio de Microbiologia Y Enfermadades Infecciosas, Madrid
- Huddinge University Hospital, Dept. of Transplantation Surgery/Immunology, Huddinge, Sweden
- United Kingdom (3):
  - Royal Free Hospital, Dept. of Haematological Oncology, London
  - Christie Hospital NHS Trust, Manchester
  - Royal Marsden Hospital, Sutton Surrey

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=60